CLINICAL TRIAL: NCT05394740
Title: A Phase Ib/II Study of Regorafenib and Nivolumab Plus Chemotherapy in Patients With Unresectable Advanced/Recurrent Gastric/Gastroesophageal Junction/Esophageal Adenocarcinoma
Brief Title: Clinical Study of Regorafenib and Nivolumab Plus Chemotherapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Principal Investigator, Kohei Shitara, Chief of Gastroenterology and Gastrointestinal Oncology Division, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC2104
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Regorafenib; Nivolumab; CapeOX; FOLFOX
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — regorafenib; Nivolumab; XELOX; Capecitabine; Oxaliplatin; Folfox protocol; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib, Nivolumab+CapeOX/FOLFOX (Experimental): Regorafenib and Nivolumab+CapeOX (Cohort A) / Nivolumab+FOLFOX (Cohort B)
  Interventions: Drug: Regorafenib; Drug: Nivolumab; Drug: CapeOX; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Regorafenib — 90 mg administered orally, once daily for 21 consecutive days followed by 7 days off
  *Repeat every 4 weeks as Regorafenib therapy
  Other Names: Stivarga
Drug: Nivolumab — CohotA:360 mg administered intravenously, every 3 weeks *Administered on the same day as CapeOX therapy Cohort B: 240 mg administered intravenously, every 2 weeks *Administered on the same day as FOLFOX therapy
  Other Names: Opdivo
Drug: CapeOX — For Cohort A only
  * Capecitabine 1,000 mg/m^2 administered orally, twice daily (Days 1 to 14 continuous dosing of CapeOX therapy)
  * Oxaliplatin 130 mg/m^2 administered intravenously (Day 1 of CapeOX therapy) *Repeat every 3 weeks as CapeOX therapy
  Other Names: XELOX; Capecitabine and Oxaliplatin
Drug: FOLFOX regimen — For Cohort B only
  * Leucovorin 400 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy)
  * Fluorouracil 400 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy) and 1,200 mg/m2 administered intravenously (Days 1 to 2 of FOLFOX therapy)
  * Oxaliplatin 85 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy) *Repeat every 2 weeks as FOLFOX therapy
  Other Names: Leucovorin, Fluorouracil and Oxaliplatin

SUMMARY:
This is an open-label, single-arm, single-center Phase Ib/II study to exploratorily evaluate the tolerability, safety, and efficacy of regorafenib and nivolumab plus chemotherapy in patients with unresectable advanced/recurrent gastric/ gastroesophageal junction/esophageal adenocarcinoma.

DETAILED DESCRIPTION:
Phase Ib part: To evaluate safety and tolerability in combination of Regorafenib, Nivolumab and chemotherapy in patient with unresectable advanced/recurrent gastric/ gastroesophageal junction/esophageal adenocarcinoma and to determine recommended dose in phase II part.

Phase II part: To evaluate safety and potential efficacy in combination of Regorafenib, Nivolumab and chemotherapy in patients in expanded arm.

The protocol treatment in this study is regorafenib and nivolumab plus CapeOX (Cohort A) / FOLFOX (Cohort B).

Regorafenib (the initial dose is 90 mg/dose) is orally administered daily for 21 days, followed by a 7-day washout period. Nivolumab is administered intravenously at a dose of 360 mg every 3 weeks (Cohort A) or 240 mg every 2 weeks (Cohort B).

Cohort A:CapeOX

* Capecitabine 1,000 mg/m^2 administered orally, twice daily (Days 1 to 14 continuous dosing of CapeOX therapy)
* Oxaliplatin 130 mg/m^2 administered intravenously (Day 1 of CapeOX therapy) *Repeat every 3 weeks as CapeOX therapy

Cohort B:FOLFOX

* Leucovorin 400 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy)
* Fluorouracil 400 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy) and 1,200 mg/m2 administered intravenously (Days 1 to 2 of FOLFOX therapy)
* Oxaliplatin 85 mg/m^2 administered intravenously (Day 1 of FOLFOX therapy) *Repeat every 2 weeks as FOLFOX therapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric/ gastroesophageal junction/esophageal adenocarcinoma that is confirmed to be unresectable/recurrent disease
2. At least 1 measurable lesion as defined by RECIST guideline version 1.1.
3. Age >= 20 years on the day informed consent is obtained
4. ECOG Performance status (PS) 0 or 1
5. The most recent laboratory value within 14 days prior to enrollment meets all of the following. (Examinations on the same day of the week 2 weeks prior to the day of enrollment may be utilized.) 1)Neutrophils >= 1,200/mm^3 2)Hemoglobin >= 8.0 g/dL 3)Platelets >= 75,000/mm^3 4)Total bilirubin <= 1.5 mg/dL 5)AST (GOT) <= 100 IU/L If liver metastases are present: <= 200 IU/L 6)ALT (GPT) <= 100 IU/L If liver metastases are present: <= 200 IU/L 7)Creatinine <= 1.5 mg/dL 8)Urine protein: any of the following (if any of the test criteria are met, other tests may not be performed.) (i)Urine protein (dipstick) <= 2+ (ii)Urine protein creatinine (UPC) ratio < 3.5 (iii)Urine protein <= 3,500 mg for 24-hour collection sample 9)PT-INR: <= 1.5 (<= 3.0 if on an anticoagulant)
6. No transfusions within 7 days prior to enrollment. (Transfusions on the same day of the week prior to enrollment are allowed)
7. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment. Both men and women must agree to use adequate contraception from the time of signing the informed consent form for a period of time (9 months in women and 7 months in men) after the last dose of protocol therapy
8. Oral administration is feasible
9. Written informed consent to participate in the study has been obtained from the patient themselves

Exclusion Criteria:

1. Prior chemotherapy for unresectable advanced/recurrent gastric/ gastroesophageal junction/esophageal adenocarcinoma (Note: Prior neoadjuvant or adjuvant therapy is allowed. However, treatment must have been completed at least 6 months prior to enrollment and progression must have occurred at least 6 months after the completion of the therapy)
2. HER2 positive (IHC3+, or IHC2+ and FISH positive)
3. Patients with hypertension that is difficult to control (systolic blood pressure >= 160 mmHg or diastolic blood pressure >= 90 mmHg) despite multiple antihypertensive medications
4. Patients with a history of acute coronary syndrome (including myocardial infarction and unstable angina), coronary angioplasty, or stent placement within 6 months prior to enrollment
5. Patients with a history or evidence of congestive heart failure of Class III or higher according to the New York Heart Association (NYHA) classification
6. Confirmed metastases to the central nervous system (Confirmation by brain computed tomography scan or magnetic resonance imaging is required at screening only if metastases to the central nervous system are clinically suspected)
7. Active double cancers with intensive treatments and possibly affect continuation of protocol treatment
8. Those with serious (needing inpatient care) complications (intestinal paralysis, intestinal obstruction, pulmonary fibrosis, poorly controlled diabetes mellitus, cardiac failure, myocardial infarction, angina pectoris, renal failure, hepatic failure, psychiatric disease, cerebrovascular disorder, ulcers requiring blood transfusions, etc.)
9. Those with active hepatitis

   * HBs antigen positive
   * HBs antibody or HBc antibody positive and HBV-DNA positive
   * Active hepatitis C (e.g., qualitative detection of HCV RNA) However, those who are HBs antigen positive may be considered eligible if HBV DNA is <1.3 log IU/mL (<2.1 log copies/mL) after treatment with antiviral drugs, such as nucleoside analogs.
10. Confirmed HIV infection
11. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease. Patients with type 1 diabetes mellitus, hypothyroidism which is manageable by hormone replacement, or skin disorders not requiring systemic treatment (such as vitiligo, psoriasis, or alopecia) are permitted to be enrolled.
12. Patients who require treatment with systemic corticosteroids (excluding temporary use for testing or prophylactic administration for allergic reactions, or for reduction of edema associated with radiotherapy), or immunosuppressants, or those treated with any of these therapies within 2 weeks prior to study enrollment
13. Patients who fail to use adequate contraception during the study participation and contraception period
14. Those unwilling or unable to comply with the protocol
15. Those considered by the principal investigator or sub-investigator as ineligible for this investigator-initiated trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs in Phase Ib part | 4weeks
  The incidence of DLTs in each cohort will be calculated for the DLT evaluable population.
ORR in Phase II part | 1 year
  ORR is defined as the proportion of subjects whose best overall response based on the RECIST guideline version 1.1 is either CR or PR.

SECONDARY OUTCOMES:
PFS | 1 year
  Progression-free survival is defined as the time from the enrollment date until the date when disease progression is determined or until the date of death from any cause, whichever comes earlier.
DoR | 1 year
  DoR is defined in responders as the period from the date of the first determination of overall response as CR or PR according to the RECIST guideline version 1.1 to the date of determination of progression (PD based on diagnostic imaging) or the date of death from any cause, whichever comes first.
DCR | 1 year
  DCR is defined as the proportion of patients in whom the best overall response was determined as CR or PR, or patients who maintained SD for 6 weeks or more according to the RECIST guideline version 1.1.
OS | 2 years
  The period will be from the day of enrollment, as the starting date of the computation, to the day of death of any cause.
Incidence of adverse events | up to 30 days after the last dose
  The treatment-emergent AEs will be summarized by CTCAE v5.0

OTHER OUTCOMES:
Biomarkers in the PhIb and PhII cohort | 1 year
  Change of ctDNA and examination of various biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Kohei Shitara, MD, Principal Investigator — National Cancer Center Hospital East
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No